CLINICAL TRIAL: NCT02254109
Title: A Randomised, Double-blind, Placebo-controlled (Within Dose Groups) Study to Evaluate Safety, Tolerability and Pharmacokinetics of Multiple Rising Inhalative Doses (50 μg, 100 μg and 200 μg q.d. for 14 Days) of BEA 2180 BR in Japanese Healthy Male Volunteers
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics of Multiple Rising of BEA 2180 BR in Japanese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1205.18
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (2):
- BEA 2180 BR - rising dose (Experimental)
  Interventions: Drug: BEA 2180 BR - rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BEA 2180 BR - rising dose
  Arms: BEA 2180 BR - rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to evaluate safety, tolerability, and pharmacokinetics of BEA 2180 BR in Japanese healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese men:

   According to the results of a complete medical history, the physical examination, vital signs (blood pressure and pulse rate), 12-lead ECG, clinical laboratory tests
2. Age ≥20 and ≤35 years
3. Body mass index (BMI) ≥18.5 and ≤25 kg/m2
4. Subjects must be able to inhale medication in a competent manner from the Respimat®
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP)

Exclusion Criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity including allergy to drug or its excipients
9. Intake of drugs with a long half-life (>24 hours) within one month or less than 10 half-lives of the respective drug before drug administration or during the trial
10. Use of prescription or non-prescription drugs within 10 days before drug Administration or during the trial. However, over-the-counter (OTC) drugs for external application (such as lubricant eye drops for contact lens, insect bite reliever) shall be allowed
11. Participation in another trial with an investigational drug within four months before drug administration or during the trial
12. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
13. Inability to refrain from smoking during the trial
14. Alcohol abuse (≥60 g/day: corresponds to ca. 3 large bottles of beer, 3 gous (ca. 540 cc) of Japanese sake, 6 shots of whisky, 6 glasses of wine or 6 glasses of Japanese shochu, distilled alcoholic beverage)
15. Drug abuse
16. Blood donation (≥100 mL within four weeks before drug administration or during the trial)
17. Excessive physical activities (within one week before drug administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site

    Exclusion criteria specific for this study:
20. Occupational (professional) exposure to antimuscarinic substances (e.g., physician, nurse, pharmacist etc.; volunteers working for medical institutions, research institutions or herb gardens)
21. History of glaucoma, urination difficulty (due to prostatic hyperplasia etc.)

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal findings in physical examination | up to 28 days after last dose administration
Number of subjects with clinically significant changes in vital signs | up to 28 days after last dose administration
  Blood pressure and pulse rate
Number of subjects with clinically significant changes in 12-lead electrocardiogram (ECG) | up to 28 days after last dose administration
Number of subjects with abnormal changes in laboratory parameters | up to 28 days after last dose administration
Number of subjects with adverse events | up to 28 days after last dose administration
Assessment of tolerability by the investigator on a 4-point scale | 28 days after last dose administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 648:00 hours
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | up to 648:00 hours
AUCτ (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ) | up to 648:00 hours
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable concentration at tz) | up to 648:00 hours
Aeτ (amount of analyte that is eliminated in urine over a uniform dosing interval τ) | up to 648:00 hours
feτ (fraction of analyte eliminated in urine over a uniform dosing interval τ) | up to 648:00 hours
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 648:00 hours
Cmin,ss (minimum concentration of the analyte in plasma at steady state) | up to 648:00 hours
Cpre,ss (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose) | up to 648:00 hours
λz,ss (terminal rate constant in plasma at steady state) | up to 648:00 hours
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | up to 648:00 hours
MRTih,ss (mean residence time of the analyte in the body at steady state after inhalation administration) | up to 648:00 hours
CL/F,ss (apparent clearance of the analyte in the plasma at steady state following extravascular multiple dose administration) | up to 648:00 hours
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | up to 648:00 hours
Accumulation ratio of the analyte in plasma based on Cmax (RA,Cmax) | up to 648:00 hours
Accumulation ratio of the analyte in plasma based on AUC (RA,AUC) | up to 648:00 hours
Accumulation ratio of the analyte in plasma based on Ae (RA,Ae) | up to 648:00 hours